CLINICAL TRIAL: NCT00110188
Title: A Phase II Study of the Efficacy and Safety of AP23573 in Patients With Taxane-Resistant Androgen-Independent Prostate Cancer (AIPC)
Brief Title: Ridaforolimus (AP23573/MK-8669) in Participants With Taxane-Resistant Androgen-Independent Prostate Cancer (AIPC)(MK-8669-017)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-017; AP23573-04-204 (Other: ARIAD protocol number)
Record Dates: First submitted 2005-05-04; First posted 2005-05-05 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — ridaforolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ridaforolimus (Experimental): 50 mg of ridaforolimis intravenously over 30 minutes, weekly
  Interventions: Drug: ridaforolimus

INTERVENTIONS:
Drug: ridaforolimus
  Other Names: deforolimus; AP23573; MK-8669; ridaforolimus was also known as deforolimus until May 2009

SUMMARY:
The purpose of this study is to assess the antitumor activity of weekly ridaforolimus study treatment in participants with taxane-resistant AIPC.

DETAILED DESCRIPTION:
The primary objective of this phase II study is to assess the anti-cancer activity of weekly ridaforolimus administration in participants with taxane-resistant AIPC. Other objectives include evaluating experimental parameters that may predict or indicate response to mTOR inhibition, such as effects on plasma VEGF, markers of tumoral PI3K/mTOR-pathway activity, and proteomic analysis. The inclusion of these evaluations in this trial may provide insight into the identification of markers that may be helpful in optimizing ridaforolimus treatment and in identifying patients with ridaforolimus-sensitive tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged ≥ 18 years with histologically documented adenocarcinoma of the prostate.
* Clinically refractory to hormone therapy (orchiectomy or luteinizing hormone-releasing hormone agonist/antagonist).
* Presence of metastatic prostate cancer that fulfills at least one evaluation category as listed: * Measurable Disease: Lesion(s) that can be accurately measured in at least one dimension with the longest diameter ≥ 20 mm using conventional techniques or ≥ 10 mm with spiral CT scan (or otherwise at least twice the reconstruction interval for CT or MRI scans). *Non-measurable disease: Lesions noted on imaging studies (including metastatic bone lesions on bone scan) or other non-measurable lesions as defined by the modified RECIST criteria. *Progressive disease following a cytotoxic chemotherapy regimen for prostate cancer.
* Previous treatment with at least one taxane-containing chemotherapy regimen. Patients may have received treatment with not more than 3 additional regimens of cytotoxic chemotherapy prior to study entry.
* Orchiectomy, or castrate levels of testosterone maintained by LHRH agonist/antagonist < 50 ng/mL.
* Predicted life expectancy > 12 weeks.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 2.
* Adequate renal and hepatic function, defined as: *Total serum bilirubin ≤ 1.5 x ULN for the institution; *AST and/or ALT ≤ 3 x ULN for the institution (≤ 5 x ULN if liver metastases are present); *Serum albumin ≥ 2.5 g/dL; *Serum creatinine ≤1.5 x ULN for the institution (or a calculated creatinine clearance ≥ 50 mL/min/1.73m2)
* Adequate bone marrow function, defined as: *ANC ≥ 1.5 x 10^9/L; *Platelet count ≥ 100 x 10^9/L
* Serum cholesterol < 350 mg/dL and triglycerides < 400 mg/dL.
* Male patients who are not surgically sterile must agree to use reliable methods of birth control for the duration of the study until 30 days after the last dose of study drug.
* Able to understand and give written informed consent.

Exclusion Criteria:

* Presence of active or progressive brain metastases.
* Prior therapy with rapamycin, rapamycin analogues or tacrolimus.
* Prior non-hormonal anticancer treatment (chemotherapy, radiotherapy, immunotherapy, biological response modifiers, signal transduction inhibitors, etc.) within 4 weeks prior to the first dose of ridaforolimus
* Ongoing toxicity associated with prior anticancer therapy (except peripheral neuropathy of ≤ grade 1 by NCI toxicity criteria).
* Another primary malignancy within the past three years (except for non-melanoma skin cancer).
* Known or suspected hypersensitivity to drugs formulated with polysorbate 80 (Tween) or any other excipient contained in the study drug.
* Known Grade 3 or 4 hypersensitivity to macrolide antibiotics (e.g., clarithromycin, erythromycin, azithromycin).
* Significant uncontrolled cardiovascular disease.
* Active infection requiring systemic therapy.
* Known HIV infection.
* Treatment with any investigational agent within 4 weeks prior to the first dose of ridaforolimus
* Concurrent treatment with immunosuppressive agents other than prescribed corticosteroids at stable doses for ≥ 2 weeks prior to first planned dose of study drug.
* Inadequate recovery from any prior surgical procedure or having undergone any major surgical procedure within 2 weeks prior to the first dose of ridaforolimus
* Presence of any other life-threatening illness or organ system dysfunction which, in the opinion of the Investigator, would either compromise the patient's safety or interfere with evaluating the safety of the study drug.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-05; Primary Completion 2007-04 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Best Overall Response (BOR) per Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 24 months

SECONDARY OUTCOMES:
Number of Participants Experiencing at Least One Adverse Event | Up to 25 months
Change from Baseline in Prostate-Specific Antigen (PSA) | Baseline and up to 24 months
Time to Tumor Progression (TTP) | Up to 24 months
Progression-Free Survival (PFS) | Up to 24 months
Overall Survival (OS) | Up to 24 months
Duration of Response (DOR) | Up to 24 months
Change from Baseline in Functional Assessment of Cancer Therapy - Prostate (FACT-P) Score | Baseline and up to 24 months
Change from Baseline in Plasma Vascular Endothelial Growth Factor (VEGF) | Baseline and Day 28 of Cycles 1 and 2 (Up to 56 days)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Haluska, M.D., Study Director — Ariad Pharmaceuticals
Locations (4):
- United States (4):
  - Louis Warchaw Prostate Cancer Center, Cedars-Sinai Medical Center, Los Angeles, California
  - Beth Israel Deaconess Medical Center/MGH/DFCI, Boston, Massachusetts
  - The Methodist Hospital Research Institute, Houston, Texas
  - University of Wisconsin, Madison, WI, Madison, Wisconsin

REFERENCES:
- [Derived] Amato RJ, Wilding G, Bubley G, Loewy J, Haluska F, Gross ME. Safety and preliminary efficacy analysis of the mTOR inhibitor ridaforolimus in patients with taxane-treated, castration-resistant prostate cancer. Clin Genitourin Cancer. 2012 Dec;10(4):232-8. doi: 10.1016/j.clgc.2012.05.001. Epub 2012 Jun 12. PMID 22695254